CLINICAL TRIAL: NCT01811979
Title: Efficacy of Oral Sucrose and Topical Anesthetics to Reduce Pain During Eye Examination
Brief Title: Efficacy of Oral Sucrose and Topical Anesthetics to Reduce Pain During Eye Examination for Retinopathy of Prematurity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Sami Ulus Children's Hospital (Other)
Responsible Party: Principal Investigator, Dilek Dilli, Assoc Prof, Dr. Sami Ulus Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 69/04.01.2012
Record Dates: First submitted 2013-03-13; First posted 2013-03-15 (Estimated); Last update posted 2013-05-09 (Estimated); Status verified 2013-05

CONDITIONS: Investigate the Efficacy of Sucrose During Eye Examination
Keywords: eye examination, oral sucrose, premature infant pain scale

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- oral sucrose solution (Active Comparator): local anesthetic eye drops (Alcaine 0.5% drop) and a pacifier, plus 0.5 cc/kg of 24% sucrose, to relieve pain associated with eye examinations for retinopathy of prematurity will be given
  Interventions: Dietary Supplement: Steril water
- steril water (Placebo Comparator): steril water 0,5 cc/kg plus topical anesthetics (Alcaine %0.5 damla) before eye examination will be given
  Interventions: Dietary Supplement: Oral sucrose solution

INTERVENTIONS:
Dietary Supplement: Oral sucrose solution — Oral sucrose solution plus topical anesthetics
  Arms: steril water
Dietary Supplement: Steril water — steril water plus topical anesthetics
  Arms: oral sucrose solution

SUMMARY:
Oral sucrose reduces pain during heel sticks and venipunctures in preterm infants. The purpose of this study was to determine the effectiveness of local anesthetic eye drops and a pacifier, plus repeated doses of 24% sucrose, to relieve pain associated with eye examinations for retinopathy of prematurity.

DETAILED DESCRIPTION:
Oral sucrose reduces pain during heel sticks and venipunctures in preterm infants. Administration of oral sucrose with and without non-nutritive sucking is the most frequently studied non-pharmacological intervention for procedural pain relief in neonates.The purpose of this study was to determine the effectiveness of local anesthetic eye drops and a pacifier, plus repeated doses of 24% sucrose, to relieve pain associated with eye examinations for retinopathy of prematurity.

ELIGIBILITY:
Inclusion Criteria:

-VLBW infants <32 weeks of gestational age

Exclusion Criteria:

* infants >32 weeks of gestational age
* neuromuscular abnormality
* major abnormality

Ages: 1 Day to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2012-04; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Premature Infant Pain Profile | two hours
  Premature Infant Pain Profile were determined after each eye examination

SECONDARY OUTCOMES:
Crying time | two hours
  Crying time will be determined after each eye examination

CONTACTS AND LOCATIONS:
Overall Officials: Eda Ç İlarslan, MD, Principal Investigator — MD
Locations (1):
- Dr Sami Ulus Children Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Stevens B, Yamada J, Lee GY, Ohlsson A. Sucrose for analgesia in newborn infants undergoing painful procedures. Cochrane Database Syst Rev. 2013 Jan 31;(1):CD001069. doi: 10.1002/14651858.CD001069.pub4. PMID 23440783
- [Derived] Dilli D, Ilarslan NE, Kabatas EU, Zenciroglu A, Simsek Y, Okumus N. Oral sucrose and non-nutritive sucking goes some way to reducing pain during retinopathy of prematurity eye examinations. Acta Paediatr. 2014 Feb;103(2):e76-9. doi: 10.1111/apa.12454. Epub 2013 Nov 11. PMID 24730361
- See also: http://www.ncbi.nlm.nih.gov/pubmed/23440783 — http://www.ncbi.nlm.nih.gov/pubmed/23440783